CLINICAL TRIAL: NCT00004055
Title: Phase II Trial of Oral Topotecan and Paclitaxel With G-CSF (Filgrastim) Support in Patients With Previously Untreated Extensive-Stage Small Cell Lung Cancer
Brief Title: Topotecan, Paclitaxel, and Filgrastim in Treating Patients With Previously Untreated Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-982052; CDR0000067251 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-12-10; First posted 2004-06-03 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Filgrastim; Paclitaxel; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- topotecan + paclitaxel + filgrastim (Experimental): Patients receive oral topotecan on days 1-5 followed by paclitaxel IV over 3 hours on day 5. Beginning 24-48 hours after chemotherapy, patients receive filgrastim (G-CSF) subcutaneously daily for up to 10 days until blood counts recover. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression. Patients who develop CNS progressive disease only should receive whole brain radiotherapy before continuing study treatment.
  Interventions: Biological: filgrastim; Drug: paclitaxel; Drug: topotecan hydrochloride

INTERVENTIONS:
Biological: filgrastim
Drug: paclitaxel
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of topotecan, paclitaxel, and filgrastim in treating patients who have previously untreated extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate oral topotecan and paclitaxel in terms of toxicity and complete and partial response rate in patients with previously untreated extensive stage small cell lung cancer. II. Determine preliminary estimates of survival in this patient population in response to this regimen.

OUTLINE: Patients receive oral topotecan on days 1-5 followed by paclitaxel IV over 3 hours on day 5. Beginning 24-48 hours after chemotherapy, patients receive filgrastim (G-CSF) subcutaneously daily for up to 10 days until blood counts recover. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression. Patients who develop CNS progressive disease only should receive whole brain radiotherapy before continuing study treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed previously untreated small cell lung cancer No mixed histology Extensive disease Metastatic disease outside the chest Contralateral supraclavicular nodes or contralateral hilar nodes outside a single radiation port OR Cytologically proven malignant pleural effusion Measurable or evaluable disease No untreated CNS metastases CNS metastases previously treated with whole brain radiotherapy allowed

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: AST no greater than 5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 5 times ULN Total bilirubin no greater than 1.5 times ULN OR Direct bilirubin normal Renal: Creatinine no greater than ULN OR Creatinine clearance at least 50 mL/min Cardiovascular: No uncontrolled angina pectoris No congestive heart failure within the past 3 months, unless ejection fraction greater than 40% No uncontrolled arrhythmias No myocardial infarction within the past 3 months Other: No significant infection No hypersensitivity to E. coli derivatives No other malignancy within the past 3 years except nonmelanoma skin cancer, carcinoma in situ of the cervix, or localized prostate cancer Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 10 years since prior chemotherapy No prior nitrosourea based chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 10 years since prior thoracic radiotherapy No more than 3 fractions of prior thoracic radiotherapy for superior vena cava syndrome Prior palliative radiotherapy except to the chest allowed No prior radiotherapy to at least 20% bone marrow No concurrent radiotherapy (including thoracic), except whole brain radiotherapy for CNS progression Surgery: At least 3 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 1999-11; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
response rate | Up to 6 months

SECONDARY OUTCOMES:
survival | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: James R. Jett, MD, Study Chair — Mayo Clinic
Locations (19):
- United States (19):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Background] Foster NR, Qi Y, Shi Q, Krook JE, Kugler JW, Jett JR, Molina JR, Schild SE, Adjei AA, Mandrekar SJ. Tumor response and progression-free survival as potential surrogate endpoints for overall survival in extensive stage small-cell lung cancer: findings on the basis of North Central Cancer Treatment Group trials. Cancer. 2011 Mar 15;117(6):1262-71. doi: 10.1002/cncr.25526. Epub 2010 Oct 19. PMID 20960500
- [Result] Molina JR, Jett JR, Foster N, Lair BS, Carroll TJ, Tazelaar HD, Hillman S, Mailliard JA, Bernath AM Jr, Nikcevich D. Phase II NCCTG trial of oral topotecan and paclitaxel with G-CSF (filgrastim) support in patients with previously untreated extensive-stage small cell lung cancer. Am J Clin Oncol. 2006 Jun;29(3):246-51. doi: 10.1097/01.coc.0000217566.11742.b5. PMID 16755177
- [Result] Jett JR, Bernath AM Jr, Hillman SL, et al.: Oral topotecan and paclitaxel with G-CSF support in patients with untreated extensive stage small cell (ED-SCLC): a phase II trial of the NCCTG. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1301, 2002.